CLINICAL TRIAL: NCT02556216
Title: Systematic Study of Parameters of Chronic Kidney Disease Mineral and Bone Disorder (CKD-MBD)
Acronym: BoneX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: University of Jena (Other)
Responsible Party: Sponsor
Other Study IDs: S 061-10.027
Record Dates: First submitted 2015-08-06; First posted 2015-09-22 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Renal Osteodystrophy
Keywords: bone biopsy; bone density
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood; urine, bone tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Bone and mineral disease is a key problem in patients with kidney disease. The available clinical parameters are non-specific, unproven for the assessment of the bone metabolism and do not reflect the complexity and diversity of the underlying bone pathology. The aim of this study is to use bone histology, novel bone markers and bone imaging results to establish a reliable decision model (diagnostic tool) that can be used to guide the individual therapy.

DETAILED DESCRIPTION:
Bone and mineral disease is a key problem in patients with kidney disease. The available clinical parameters are non-specific, unproven for the assessment of the bone metabolism and do not reflect the complexity and diversity of the underlying bone pathology.

In this study bone histology parameters including results of tetracycline labeling will be compared to non-invasive parameters of bone metabolism (e.g. sclerostin, calciprotein particles) and bone structure obtained by imaging (e.g. bone density).

The aim of the study is to establish a reliable decision model (diagnostic tool) with these non-invasive parameters that can be used to guide the individual therapy. The decision model will be based on single calculations of the area under the curve for each parameter, including determination of the optimal cutpoint, sensitivity and specificity. These results will be integrated in a multivariate logistic regression analysis. The resulting model will enable to calculate the individual probability of the underlying bone diagnosis as a single value (without a specific dimension).

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney disease who have an indication for a bone biopsy, based on clinical, laboratory and radiologic findings

Exclusion Criteria:

* known malignant bone or bone marrow disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease (including kidney transplanted patients) with mineral and bone disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of a diagnostic model (derived from the non-invasive radiologic and blood parameters of the bone) in relation to the 'gold standard' bone biopsy result | cross-sectional study, one week
  After determining the AUC, sensitivity, specificity and optimal cutpoint for each parameter, a logistic regression model is created which gives the probability of the underlying bone diagnosis as a single probability value.
  In this cross-sectional studies each patient gets a one-time assessment of radiologic and blood parameters of bone metabolism obtained within one week. Accuracy is described by the performance measures sensitivity, specificity, area under the curve, negative and positive predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Margret Patecki, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided